CLINICAL TRIAL: NCT04374214
Title: Effect of Simvastatin on Success of Pulpotomy in Cariously Exposed Permanent Molars: a Randomized Control Trial
Brief Title: Effect of Simvastatin as Pulpotomy Agent in Cariously Exposed Permanent Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr Sudeepender Gehlot
Record Dates: First submitted 2020-04-22; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Reversible Pulpitis
Keywords: Permanent teeth; Complete pulpotomy; Simvastatin -alpha tricalcium phosphate; Mineral Trioxide Aggregate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete Pulpotomy using mineral trioxide aggregate (Active Comparator): Twenty-eight patients with curiously exposed permanent molars will be treated with complete pulpotomy by using Mineral Trioxide Aggregate.
  Interventions: Procedure: Complete Pulpotomy using Mineral Trioxide Aggregate
- Complete Pulpotomy using Simvastatin-alphatricalcium phosphate (Active Comparator): Twenty-eight patients with curiously exposed permanent molars will be treated with complete pulpotomy by using Simvastatin -alphatricalcium phospahte.
  Interventions: Procedure: Complete Pulpotomy using Simvastain -alphatricalcium phosphate

INTERVENTIONS:
Procedure: Complete Pulpotomy using Mineral Trioxide Aggregate — Inflammed coronal pulp tissue will be removed till the canal orifices and mineral trioxide aggregate placed over the amputated pulp stump.
  Arms: Complete Pulpotomy using mineral trioxide aggregate
Procedure: Complete Pulpotomy using Simvastain -alphatricalcium phosphate — Inflammed coronal pulp tissue will be removed till the canal orifices and Simvastatin -alpha tricalcium phosphate placed over the amputated pulp stump.
  Arms: Complete Pulpotomy using Simvastatin-alphatricalcium phosphate

SUMMARY:
The study will compare the outcome of complete pulpotomy in mature permanent mandibular molars with deep carious lesions by using Mineral Trioxide Aggregate and Simvastatin -alpha tricalcium phosphate as medicament agent

DETAILED DESCRIPTION:
After a thorough history, clinical and radiographic examination with all eligibility confirmation, written informed consent will be taken from the patient after explaining the procedure, its associated risks and benefits. Clinical diagnosis of reversible pulpitis will be established. Complete pulpotomy will be done in both groups. Mineral Trioxide Aggregate and Simvastatin -alpha tricalcium phosphate will be used as pulpotomy agents. Pain analysis will be carried out preoperatively and postoperatively at every 6 hours for 1 day and then every 24 hours till 7 days after the intervention. All the subjects will be followed up for evaluation of clinical and radiographic success at 3, 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patient willing to participate in the study.
2. Age group of 15 to 40 years
3. Mature permanent mandibular molars with reversible pulpitis (positive response on the cold test and early response as compared to the adjacent or contralateral tooth)
4. Teeth exhibiting occlusal pulp exposure from primary dental caries.
5. Absence of periapical lesions assessed by radiographic examination.
6. Tooth demonstrating no mobility or swelling and no tenderness to percussion or palpation

Exclusion Criteria:

1. Primary teeth.
2. Teeth with irreversible pulpitis (spontaneous pain) or pulp necrosis, chronic periodontitis, cracked tooth, internal or external resorption, calcified canals, associated with sinus tract and furcation or apical radiolucency.
3. Immune-compromised, pregnant and patients with any systemic disorder.
4. Patients taking statin medication.
5. Failure to obtain authorization from the patient.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success | Baseline to 12 months
  criteria for successful clinical outcome will be absence of clinical sign and symtoms which include Absence of tenderness to percussion,tooth mobility of grade 1 or less.Absence of associated soft tissue swelling or tenderness to palpation.

SECONDARY OUTCOMES:
Pain analysis | Baseline to 7 days
  Assess the incidence and intensity of pain postoperatively at every 6 hours to 1 day till 7d ays using Visual Analogue scale.Pain intensity will be noted as no pain (0-4mm), mild pain (5-44), moderate pain (45-74mm) and severe pain (75-100mm) on the scale of 0-100mm
Radiographic success | Baseline to 12 months
  Radiographic success will be evaluated by change in periapical index (PAI) scores.
  PAI score 1: Normal periapical structure PAI score 2: Small changes in bone structure PAI score 3: Changes in bone structure with some mineral loss PAI score 4: Periodontis with well defined radiolucent area PAI score 5: Severe periodontitis with elements indicating expansion of lesion

CONTACTS AND LOCATIONS:
Overall Officials: Sudeepender Gehlot, Principal Investigator — PGIDS, Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India

REFERENCES:
- [Derived] Gehlot S, Kumar V, Mittal S, Duhan J, Sangwan P, Arora M, Chauhan N. Effect of Simvastatin on Success of Pulpotomy in Carious Permanent Molars With Symptomatic Irreversible Pulpitis: A Randomised Controlled Trial. Aust Endod J. 2026 Feb 6. doi: 10.1111/aej.70062. Online ahead of print. PMID 41652862